CLINICAL TRIAL: NCT06672224
Title: Prospective Analysis of Patients at Risk for Breast Cancer-Related Lymphedema (BCRL) Using Indocyanine Green (ICG) Fluoroscopy and SPYTM Angiography
Brief Title: Indocyanine Green Fluoroscopy and SPY Angiography for the Assessment of Lymphatic Structure in Breast Cancer Patients at Risk for Breast Cancer-Related Lymphedema
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: low accrual
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 23823; NCI-2024-08855 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23823 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer-Related Lymphedema; Breast Carcinoma
MeSH Terms: conditions — Breast Cancer Lymphedema; Breast Neoplasms | interventions — Fluid Therapy; Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive Care (ICG, fluid, SPY, lymphedema assessment) (Experimental): Patients receive ICG dye SC and receive fluids IV over one hour and undergo SPY imaging and lymphedema assessment on day 1. Patients also receive ICG dye and undergo imaging and lymphedema assessments again at 1, 3, 6, and 12 months on study.
  Interventions: Procedure: Fluid Therapy; Drug: Indocyanine Green; Other: Questionnaire Administration; Other: Research or Clinical Assessment Tool; Procedure: SPY Elite Fluorescence Imaging; Other: Survey Administration

INTERVENTIONS:
Procedure: Fluid Therapy — Given IV
Drug: Indocyanine Green — Given subcutaneously
  Other Names: ICG
Other: Questionnaire Administration — Ancillary studies
Other: Research or Clinical Assessment Tool — Undergo lymphedema assessment
  Other Names: Clinical Assessment Tool; Clinical or Research Assessment Tool
Procedure: SPY Elite Fluorescence Imaging — Undergo SPY imaging
  Other Names: SPY Elite; SPY Elite Imaging
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial assesses the change in lymphatic structure from placement of an intravenous (IV) line and fluid administration using a diagnostic agent, indocyanine green (ICG), with SPY (Trademark) angiography in breast cancer patients at risk for breast cancer-related lymphedema (BCRL). Patients that are diagnosed with breast cancer with lymph node involvement often undergo treatment that includes surgery to remove the axillary nodes and radiation. Unfortunately, this procedure increases the incidence of BCRL in the surgical arm, as well as other problems including heaviness of the arm, fibrotic skin changes, and an increase in infection risk. Because of these symptoms, venipuncture (blood draw) is often avoided in these arms. Researchers want to show that placement of an IV line and fluid administration in patients at risk for BCRL will indeed not alter the lymphatic structure of the arm and will not change the incidence of BCRL by administering indocyanine green (ICG) dye to patients and assessing their arm lymphatics. ICG is a fluorescent dye that is able to be visualized by the SPY angiography imaging system as it travels through the lymphatic system, allowing researchers to assess how well blood flows throughout the body. Receiving ICG and undergoing SPY angiography may be effective in showing that placement of an IV and fluid administration in breast cancer patients at risk for BCRL will not alter the lymphatic structure of their arm and will not change the incidence of BCRL.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Assess the change in lymphatic architecture resulting from placement of an IV line and fluid administration in patients at risk for BCRL.

SECONDARY OBJECTIVES:

I. Identify changes in presence/severity of lymphedema based on:

Ia. SOZO Digital Health Platform scale; Ib. Patient self-reported outcomes; Ic. Arm circumference. II. Assess association between SOZO scale, MD Anderson Cancer Center (MDACC) lymphedema score (LS), and patient-reported outcomes.

EXPLORATORY OBJECTIVES:

I. Observe changes in mapping of superficial lymphatics that are responsible for the upper extremity arm with use of ICG dye and SPY angiography.

II. Identify risk factors associated with higher rates of lymphedema after IV line/fluid administration.

OUTLINE:

Patients receive ICG dye subcutaneously (SC) and receive fluids IV over one hour and undergo SPY imaging and lymphedema assessment on day 1. Patients also receive ICG dye and undergo imaging and lymphedema assessments again at 1, 3, 6, and 12 months on study.

ELIGIBILITY:
Inclusion Criteria:

* Documented written informed consent of the participant
* Men or women age: >= 18 years
* Diagnosis of breast cancer
* Full axillary dissection at least 12 months prior
* Patient needs vena puncture and has problem with access in the contralateral arm. Recruitment includes patients who do not wish to use their contralateral arm, lower extremities, or central access through their neck, as well as patients for whom multiple attempts result in increased anxiety, discomfort, and treatment delays
* No clinical evidence of lymphedema by MD Anderson grading system and normal SOZO values compared to contralateral arm
* Willingness to:

  * Complete Lymphedema Life Impact Scale (LLIS) survey
  * Allow measurement of arm circumference, bioimpedance, and ICG imaging in real time
  * Permit medical record/clinical laboratory result review

Exclusion Criteria:

* Patients with active malignancy (i.e., currently undergoing treatment), infection, or bleeding tendency
* Diagnosis of lymphedema
* Women of childbearing potential: pregnant/nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-08-14 (Estimated); Primary Completion 2026-08-14 (Estimated); Study Completion 2026-08-14 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with worsening lymphedema in the affected arm | Baseline to 12 months
  Measured by the MD Anderson Cancer Center (MDACC) lymphedema score (LS) (measured on a scale of 0 to 5) increased by at least 1 level. Will be estimated as a percentage of patients with MDACC lymphedema score that is at least 1 unit worse at 12 months than at baseline; 95% confidence interval (CI) will be calculated.

SECONDARY OUTCOMES:
Change in lymphedema severity based on SOZO Digital Health Platform scale | Baseline to 12 months
  Will be calculated (with appropriate confidence intervals); Pearson (or Spearman, as appropriate) correlation coefficients will be calculated to assess the strength of relationship between all four assessment methods (all time points). Graphical representation of data will be used to help understand and assess the nature of the relationship of these modalities.
Change in patient self-reported outcomes scores | Baseline to 12 months
  Will be calculated (with appropriate confidence intervals); Pearson (or Spearman, as appropriate) correlation coefficients will be calculated to assess the strength of relationship between all four assessment methods (all time points). Graphical representation of data will be used to help understand and assess the nature of the relationship of these modalities.
Change in arm circumference measurements | Baseline to 12 months
  Will be calculated (with appropriate confidence intervals); Pearson (or Spearman, as appropriate) correlation coefficients will be calculated to assess the strength of relationship between all four assessment methods (all time points). Graphical representation of data will be used to help understand and assess the nature of the relationship of these modalities.
Correlation between lymphedema assessment methods (1) MDACC LS, (2) patient-reported outcomes, (3) SOZO scale, and (4) arm circumference | Baseline to 12 months
  Will be calculated (with appropriate confidence intervals); Pearson (or Spearman, as appropriate) correlation coefficients will be calculated to assess the strength of relationship between all four assessment methods (all time points). Graphical representation of data will be used to help understand and assess the nature of the relationship of these modalities.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Chang, Principal Investigator — City of Hope Medical Center